CLINICAL TRIAL: NCT01007591
Title: Calcipotriol Plus Hydrocortisone in Paediatric Patients (Aged 6 to 17 Years) With Psoriasis Vulgaris on the Face and on the Intertriginous Areas
Brief Title: A Study Comparing LEO 80190 Ointment With Hydrocortisone Ointment, Both Applied Once Daily in the Treatment of Psoriasis Vulgaris on the Face and Intertriginous Areas
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: LEO Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LEO 80190-O25
Record Dates: First submitted 2009-11-03; First posted 2009-11-04 (Estimated); Results first posted 2019-01-15 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2018-03

CONDITIONS: Psoriasis Vulgaris
MeSH Terms: interventions — Hydrocortisone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- LEO 80190 ointment (Active Comparator)
  Interventions: Drug: LEO 80190
- Hydrocortisone 10 mg/g ointment (Active Comparator)
  Interventions: Drug: Hydrocortisone

INTERVENTIONS:
Drug: LEO 80190 — Applied once daily
  Arms: LEO 80190 ointment
Drug: Hydrocortisone — Applied once daily
  Arms: Hydrocortisone 10 mg/g ointment

SUMMARY:
An international, multi-centre, prospective, randomised, double-blind, active-controlled, 2-arm, parallel group, 8-week, phase 3 clinical study in paediatric patients (aged 6 to 17 years) with psoriasis vulgaris on the face and on the intertriginous areas

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of psoriasis vulgaris involving the face
* Clinical signs of psoriasis vulgaris on the trunk and/or on the limbs, or earlier diagnosed with psoriasis vulgaris on the trunk and/or limbs. The extent and severity of psoriasis vulgaris on trunk and/or limbs should be amenable to topical therapy with any of the allowed medications
* An extent of psoriatic involvement of the face of at least 5 cm2 (the sum of all facial lesions)
* Treatment areas (the face and the intertriginous areas) amenable to topical treatment with a maximum of 30 g (6 to 11 years) or 45 g (12 to 17 years) of ointment per week
* Disease severity graded as mild, moderate or severe according to the investigator's global assessment of disease severity of the face
* Aged 6 to 17 years

Exclusion Criteria:

* Systemic treatment with therapies other than biologicals with a potential effect on psoriasis vulgaris within the 4-week period prior to randomisation
* Systemic treatment with biological therapies (marketed or not marketed) with a possible effect on psoriasis vulgaris within 4 weeks (etanercept), 2 months (adalimumab, alefacept, infliximab), 4 months (ustekinumab) or 4 weeks/5 half-lives (which-ever is longer) for experimental biological products prior to randomisation
* PUVA therapy or Grenz ray therapy within the 4-week period prior to randomisation
* UVB therapy within the 2-week period prior to randomisation
* Topical treatment of psoriasis vulgaris lesions on the face or on the intertriginous areas within the 2-week period prior to randomisation
* Topical treatment with very potent WHO group IV corticosteroids within the 2-week period prior to randomisation
* Initiation of or expected changes to concomitant medication that may affect psoriasis vulgaris (e.g., beta blockers, anti-malaria drugs, lithium and ACE inhibitors) during the treatment phase of the study
* Current diagnosis of erythrodermic, exfoliative or pustular psoriasis

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2009-10; Primary Completion 2010-06 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Frédéric Cambazard, MD, Principal Investigator — FRANCE
Locations (1):
- CHU Saint-Etienne Hôpital NOrd, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | LEO 80190 Ointment | Hydrocortisone 10 mg/g Ointment
Started | 27 | 13
Completed | 26 | 12
Not Completed | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | LEO 80190 Ointment | Hydrocortisone 10 mg/g Ointment | Total
Number analyzed (Participants) | 27 | 13 | 40
Age, Customized [Count of Participants; unit: Participants]
  Years: 6-8 | 6 | 3 | 9
  Years: 9-11 | 8 | 4 | 12
  Years: 12-14 | 5 | 2 | 7
  Years: 15-17 | 8 | 4 | 12
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 7 | 26
  Male | 8 | 6 | 14
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 6 | 2 | 8
  France | 10 | 6 | 16
  Germany | 11 | 5 | 16

OUTCOME MEASURES:

1. Primary Outcome: The Percentage Change in Psoriasis Area and Severity Index (PASI) of the Face Last Observation Carried Forward (LOCF) at End of Treatment
Description: PASI of the face was to be calculated based on the (sub)investigator's assessment of extent (E), redness (R), thickness (T) and scaliness (S) using the following formula:
  0.05 (R+T+S) E
  It ranged from 0 to 3.6.
Time Frame: From baseline (Day 0) to end of treatment (Week 8)
Measure: Mean (Standard Deviation); unit: percentage of change in PASI
Arm/Group | LEO 80190 Ointment | Hydrocortisone 10 mg/g Ointment
Number analyzed (Participants) | 27 | 13
percentage of change in PASI | -60.8 (51.1) | -54.2 (59.2)
Statistical Analysis 1: Comparison: LEO 80190 Ointment vs Hydrocortisone 10 mg/g Ointment; Test type: Superiority; p = 0.75, ANOVA; Treatment comparison using an ANOVA model with age group and treatment as design variables; Mean Difference (Final Values) = -6.02, 95% CI 2-sided [-43.7 to 31.7]

2. Secondary Outcome: Participants With "Controlled Disease" According to the Investigator's Global Assessment (IGA) of Disease Severity on the Face LOCF
Description: For subjects with a baseline (Day 0) severity of moderate or worse - "controlled disease" of the face was defined as clear or almost clear according to the IGA of the face.
  For subjects with a baseline (Day 0) severity of mild - "controlled disease" of the face was defined as clear according to the IGA of the face.
  At baseline (Day 0) to end of treatment (Week 8) the (sub) investigator made an assessment of the disease severity of the face using the 6-category scale below.
  Clear, almost clear, mild, moderate, severe and very severe.
Time Frame: At end of treatment (Week 8)
Measure: Count of Participants; unit: Participants
Arm/Group | LEO 80190 Ointment | Hydrocortisone 10 mg/g Ointment
Number analyzed (Participants) | 27 | 13
Participants
  Controlled | 13 | 7
  Non-controlled | 14 | 6

3. Secondary Outcome: The Percentage Change in PASI of the Face LOCF at Week 4
Description: as for outcome 1
Time Frame: From baseline (Day 0) to Week 4 (Day 28)
Measure: Mean (Standard Deviation); unit: percentage of change in PASI
Arm/Group | LEO 80190 Ointment | Hydrocortisone 10 mg/g Ointment
Number analyzed (Participants) | 27 | 13
percentage of change in PASI | -54.8 (33.8) | -54.9 (37.3)

4. Secondary Outcome: Participants With "Controlled Disease" According to the Investigator's Global Assessment (IGA) of Disease Severity of the Intertriginous Areas LOCF
Description: At baseline (Day 0) to end of treatment (Week 8) the (sub)investigator made an assessment of the disease severity of the intertriginous areas using the following 6-category scale.
  Clear, almost clear, mild, moderate, severe and very severe.
  For subjects with a baseline (Day 0) severity of moderate or worse - "controlled disease" of the intertriginous areas was defined as clear or almost clear according to the IGA of the intertriginous areas.
  For subjects with a baseline (Day 0) severity of mild - "controlled disease" of the intertriginous areas was defined as clear according to the IGA of the intertriginous areas.
Time Frame: At end of treatment (Week 8)
Population: The intertriginous analysis set consisted of all participants having 'Mild' or worse according to IGA of the intertriginous areas at baseline. The intertriginous analysis set therefore consisted of 11 participants.
Measure: Count of Participants; unit: Participants
Arm/Group | LEO 80190 Ointment | Hydrocortisone 10 mg/g Ointment
Number analyzed (Participants) | 7 | 4
Participants
  Controlled | 2 | 4
  Non-controlled | 5 | 0

5. Secondary Outcome: The Percentage Change in Total Sign Score (TSS) of the Intertriginous Areas LOCF
Description: For each clinical sign, a single score, reflecting the average severity of all psoriatic lesions on the intertriginous areas was determined according to the scale below:
  Redness 0.none
  1. mild
  2. moderate
  3. severe
  4. very severe
  Thickness
  0.none
  1. mild
  2. moderate
  3. severe
  4. very severe
  Scaliness
  0.none
  1. mild
  2. moderate
  3. severe
  4. very severe A mean score was calculated for each sign (redness, thickness and scaliness) based on scores of all the defined intertriginous areas with psoriasis at baseline and the sum of these mean scores constituted the TSS ranging from 0 to 12.
Time Frame: From baseline (Day 0) to end of treatment (Week 8)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: percentage in TSS
Arm/Group | LEO 80190 Ointment | Hydrocortisone 10 mg/g Ointment
Number analyzed (Participants) | 7 | 4
percentage in TSS | -56.6 (38.2) | -93.2 (8.2)

ADVERSE EVENTS:
Time Frame: From baseline (Day 0) to follow-up
Description: Follow-up visit only applicable if an AE (serious or non-serious) classified as possibly / probably related to the study medication or not assessable in relation to the study medication was present at the subject's last on-treatment visit. This follow-up had to be performed 14 ± 2 days after the subject's last on-treatment visit or until final outcome of the AE was determined, whichever came first.
Arm/Group | LEO 80190 Ointment | Hydrocortisone 10 mg/g Ointment
All-Cause Mortality (participants affected / at risk) | 0/27 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/13
Other Adverse Events (participants affected / at risk) | 17/27 | 9/13
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | LEO 80190 Ointment (N=27) | Hydrocortisone 10 mg/g Ointment (N=13)
Ear pain (Ear and labyrinth disorders) | 1 | 0
Conjunctivitis (Eye disorders) | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 2 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0
Application site burning (General disorders) | 1 | 0
Influenza like illness (General disorders) | 1 | 0
Pyrexia (General disorders) | 1 | 0
Acute tonsillitis (Infections and infestations) | 1 | 0
Bladder infection (Infections and infestations) | 1 | 0
Bronchitis (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 2 | 0
Herpes simplex (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 1 | 2
Nasopharyngitis (Infections and infestations) | 5 | 2
Pharyngitis streptococcal (Infections and infestations) | 1 | 0
Tonsillitis (Infections and infestations) | 1 | 0
Joint sprain (Injury, poisoning and procedural complications) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Headache (Nervous system disorders) | 3 | 1
Dysmenorrhoea (Reproductive system and breast disorders) | 1 | 0
Pruritus genital (Reproductive system and breast disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Erythema (Skin and subcutaneous tissue disorders) | 2 | 0
Nail dystrophy (Skin and subcutaneous tissue disorders) | 1 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 3 | 0
Rash scaly (Skin and subcutaneous tissue disorders) | 1 | 0
Skin burning sensation (Skin and subcutaneous tissue disorders) | 1 | 0
Skin irritation (Skin and subcutaneous tissue disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Company acknowledges the investigators' right to publish the entire results of the study, irrespective of outcome. The Company retains the right to have any publication submitted to the Company for review at least 30 days prior to the same paper being submitted for publication or presentation. Investigators must undertake not to submit any part of their individual data for publication without the prior consent of LEO.